CLINICAL TRIAL: NCT03716752
Title: Modified Connective Tissue Graft Wall With Wing Technique for Posterior Teeth in Treating One Wall Vertical Bone Defects With Class III Gingival Recession: A 12 Months Follow up
Brief Title: Modified Connective Tissue Graft Wall With Wing Technique for Posterior Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, nermin mohammed ahmed yussif, assistant lecturer, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1235
Record Dates: First submitted 2018-10-13; First posted 2018-10-23 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Recession
Keywords: connective tissue wall technique; modified connective tissue wall technique with a wing; recession defects in posterior teeth; recession defects with infrabony defects
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bone graft and collagen barrier (Active Comparator): peridoontal regeneration using bone graft and collagen barrier as treatment of vertical bony defects with recession defect
  Interventions: Procedure: Modified connective tissue graft wall with wing technique
- Modified connective tissue graft wall with wing technique (Experimental): peridoontal regeneration using bone graft and modified connective tissue graft wall with wing as treatment of vertical bony defects with recession defect
  Interventions: Procedure: Modified connective tissue graft wall with wing technique

INTERVENTIONS:
Procedure: Modified connective tissue graft wall with wing technique — the usage of bone graft and collagen barrier to treat recession defects accompanied vertical bony defcets in posterior teeth
  Other Names: bone graft and collagen barrier

SUMMARY:
The investigators reported here the application of usage modified connective tissue graft wall technique for posterior teeth. The treatment outcomes suggested the efficacy of the used technique in treating recession defects accompanied by infrabony defects in molars.

DETAILED DESCRIPTION:
Gingival recession is defined as the apical migration of the gingival margin leaving the root surface denuded. Treatment of Class III and IV defects and achievement good of results seems to be quite difficult due to the advanced loss of the soft and hard tissues supporting the affected teeth. Furthermore, partial to total loss of the interproximal papilla is one of the main challenges that contribute for achieving higher levels of esthetics especially in anterior zone. In such a case, conventional techniques of root coverage results usually in poor prognosis.

ELIGIBILITY:
Inclusion Criteria:

* recession defects in posterior teeth
* vertical infrabony defects in relation to the same recession defect

Exclusion Criteria:

* smokers
* suystemic diseases
* pregnency and lactating mothers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
recession defect dimensions | 12 months
  measurment of recession defect depth and width

CONTACTS AND LOCATIONS:
Locations (1):
- Octobar University of Modern Sciences and Arts, Giza, Egypt